CLINICAL TRIAL: NCT03333928
Title: A Proof-of-Concept and Dose-Ranging Study Investigating the Efficacy and Safety of HTD1801 in Adult Subjects With Primary Sclerosing Cholangitis (PSC)
Brief Title: A POC and Dose-Ranging Study of HTD1801 in PSC Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HighTide Biopharma Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HTD1801.PCT003
Record Dates: First submitted 2017-10-27; First posted 2017-11-07 (Actual); Results first posted 2022-04-06 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Primary Sclerosing Cholangitis (PSC)
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Intervention Model Description: A primary parallel group comparison for a 6-week treatment period (Period 1), followed by a 6-week dose-controlled extension (Period 2), and followed by a 6-week placebo-controlled randomized withdrawal (Period 3).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- HTD1801 500 mg BID (Active Comparator)
  Interventions: Drug: HTD1801
- HTD1801 1000 mg BID (Active Comparator)
  Interventions: Drug: HTD1801
- Placebo BID (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HTD1801 — HTD1801 tablets, 250 mg
  Arms: HTD1801 1000 mg BID; HTD1801 500 mg BID
Drug: Placebo — tablets manufactured to mimic HTD1801 tablets
  Arms: Placebo BID

SUMMARY:
The study was a dose-ranging, 18-week study comparing two doses of HTD1801 (500 mg BID and 1000 mg BID) to placebo in adult subjects with PSC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 75 years of age;
* Have a clinical diagnosis of PSC as evident by chronic cholestasis of more than six months duration with either a consistent magnetic resonance cholangiopancreatography (MRCP)/endoscopic retrograde cholangiopancreatography (ERCP) showing sclerosing cholangitis;
* If subjects have Inflammatory Bowel Disease (IBD) they will be eligible to participate. If a subject has IBD, documented evidence of IBD must have been evident by prior endoscopy or in previous medical records for ≥6 months. In addition, subjects may only enter the study with a Partial Mayo Score of 0-4, inclusively. Subjects who are on treatment are allowed, provided they are stable for 3 months if taking:

  1. 5-amino salicylic acid drugs,
  2. azathioprine,
  3. 6-mercaptopurine, or methotrexate
  4. biologics;
* Have a serum ALP ≥1.5 × upper limit of normal (ULN);
* Be able to understand and sign a written informed consent form (ICF);
* Subjects receiving allowed concomitant medications need to be on stable therapy for 28 days prior to the Baseline visit, with the exception of ursodeoxycholic acid (UDCA), which should be stable for at least 6 weeks prior to the Baseline visit.

Exclusion Criteria:

* Presence of documented secondary sclerosing cholangitis (such as ischemic cholangitis, recurrent pancreatitis, intraductal stone disease, severe bacterial cholangitis, surgical or blunt abdominal trauma, recurrent pyogenic cholangitis, choledocholithiasis, toxic sclerosing cholangitis due to chemical agents, or any other cause of secondary sclerosing cholangitis) on prior clinical investigations;
* Small duct PSC;
* Presence of percutaneous drain or bile duct stent;
* History of cholangiocarcinoma or clinical suspicion of new dominant stricture within 1 year by MRCP/ERCP. Presence of dominant stricture without ERCP evidence of cholangiocarcinoma is acceptable if stable for ≥ 1 year;
* Ascending cholangitis within 60 days prior to Screening;
* History of alcohol or substance abuse or dependence;
* Prior or planned liver transplantation;
* Presence of alternative causes of chronic liver disease, including alcoholic liver disease, nonalcoholic steatohepatitis, primary biliary cirrhosis, autoimmune hepatitis;
* Platelet count below 125,000/mm3, albumin below 3.0 g/dL, International Normalized Ratio (INR) > 1.2, or a history of ascites, or encephalopathy, or history of esophageal variceal bleeding;
* Severe active IBD or flare in colitis activity within the last 90 days requiring intensification of therapy beyond baseline treatment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Di Bisceglie, MD,FACP,FAASLD, Study Director — HighTide Therapeutics USA, LLC
Locations (26):
- United States (24):
  - Arizona Liver Health, Chandler, Arizona
  - Arizona Liver Health, Tuscon, Arizona
  - Fresno Clinical Research Center, Fresno, California
  - Keck School of Medicine of USC, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Colorado, Denver, Aurora, Colorado
  - South Denver Gastroenterology, PC, Englewood, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Florida Research Institute, Lakewood Rch, Florida
  - University of Miami, Miami, Florida
  - Mercy Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Michigan Medicine University of Michigan, Ann Arbor, Michigan
  - Gastrointestinal Associates, Flowood, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai - Icahn School of Medicine, New York, New York
  - Cumberland Research Associates, Fayetteville, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Pinnacle Clinical Research, Austin, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - Swedish Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
- Canada (2):
  - Aspen Woods Clinic, Calgary, Alberta
  - Toronto Centre for Liver Disease, Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kowdley KV, Forman L, Eksteen B, Gunn N, Sundaram V, Landis C, Harrison SA, Levy C, Liberman A, Di Bisceglie AM, Hirschfield GM. A Randomized, Dose-Finding, Proof-of-Concept Study of Berberine Ursodeoxycholate in Patients With Primary Sclerosing Cholangitis. Am J Gastroenterol. 2022 Nov 1;117(11):1805-1815. doi: 10.14309/ajg.0000000000001956. Epub 2022 Aug 22. PMID 36327436

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-nine subjects were recruited from 23 academic medical centers and community clinics in the US and Canada. The first subject was enrolled on 18 June 2018 and the last subject last visit was completed on 10 Aug 2020.
Groups:
- 500mg HTD1801 BID; 1000 mg HTD1801 BID: HTD1801: HTD1801 tablets, 250 mg
Period: Initial Dosing Period (Period 1)
Arm/Group | 500mg HTD1801 BID | 1000 mg HTD1801 BID | Placebo BID
Started | 16 | 25 | 18
Completed | 15 | 21 | 14
Not Completed | 1 | 4 | 4
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Corporate decision to not initiate dosing in new patients because of COVID-19 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 3 | 1
Period: Dose-controlled Extension (Period 2)
Arm/Group | 500mg HTD1801 BID | 1000 mg HTD1801 BID | Placebo BID
Started (Subjects randomized to active treatment remained on their Period 1 dose. Subjects who had been randomized to Placebo during Period 1 were randomized 1:1 to either HTD1801 500 mg BID or HTD1801 1000 mg BID.) | 22 | 29 | 0
Completed | 19 | 28 | 0
Not Completed | 3 | 1 | 0
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Period: Randomized Withdrawal (Period 3)
Arm/Group | 500mg HTD1801 BID | 1000 mg HTD1801 BID | Placebo BID
Started (Active subjects from Period 2 were re-randomized in Period 3 to receive either Placebo, HTD1801 500 mg BID or HTD 1000 mg BID.) | 10 | 14 | 26
Completed | 8 | 14 | 25
Not Completed | 2 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 59 subjects were randomized into the study, 55 subjects were included in the safety population and 54 subjects were included in the modified intent-to-treat population (mITT). Four subjects were randomized but did not get study drug - two subjects were not started on study drug because of COVID-19, one subject did not meet eligibility criteria and one subject withdrew consent.
Groups:
- HTD1801 500 mg BID; HTD1801 1000 mg BID: HTD1801: HTD1801 tablets, 250mg
- Total: Total of all reporting groups
Arm/Group | HTD1801 500 mg BID | HTD1801 1000 mg BID | Placebo BID | Total
Number analyzed (Participants) | 15 | 24 | 16 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (13.6) | 45 (13.7) | 40 (15.8) | 43 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 9 | 23
  Male | 11 | 14 | 7 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 2 | 7
  White | 14 | 19 | 13 | 46
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Serum Alkaline Phosphatase (ALP) From Baseline to Week 6 in Period 1
Time Frame: Baseline to Week 6
Population: Modified Intent-to-Treat (mITT) population: 59 subjects were randomized; however, 4 subjects did not receive the study drug. The remaining 55 subjects were dosed with study drug; however, 1 subject was excluded due to the absence of baseline assessments and withdrew due to AE on Day 2. The mITT population consisted of the remaining 54 subjects. Subjects were randomized to receive HTD1801 BID doses of 500 mg, 1000 mg, or matching placebo for 6 weeks.
Measure: Mean (Standard Error); unit: U/L
Arm/Group | HTD1801 500 mg BID | HTD1801 1000 mg BID | Placebo BID
Number analyzed (Participants) | 15 | 23 | 16
U/L | -71 (136.9) | -73 (139.9) | 94 (261.7)

2. Secondary Outcome: Percentage of Subjects Who Achieve ALP of <1.5 x ULN at the End of Week 6 (Period 1)
Time Frame: Baseline to Week 6
Population: Period 1 mITT population: 54 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | HTD1801 500 mg BID | HTD1801 1000 mg BID | Placebo BID
Number analyzed (Participants) | 15 | 23 | 16
Participants | 2 | 6 | 1

3. Secondary Outcome: Percentage of Subjects Who Achieve a 50% Decrease in ALP at the End of Week 6 (Period 1)
Time Frame: Baseline to Week 6
Population: Period 1 mITT population: 54 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | HTD1801 500 mg BID | HTD1801 1000 mg BID | Placebo BID
Number analyzed (Participants) | 15 | 23 | 16
Participants | 1 | 4 | 0

4. Secondary Outcome: Percentage of Subjects Who Normalize ALP at the End of Week 6 (Period 1)
Time Frame: Baseline to Week 6
Population: Period 1 mITT population: 54 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | HTD1801 500 mg BID | HTD1801 1000 mg BID | Placebo BID
Number analyzed (Participants) | 15 | 23 | 16
Participants | 0 | 2 | 0

5. Secondary Outcome: Absolute Change in Serum Total Bilirubin at the End of Week 6 (Period 1)
Time Frame: Baseline to Week 6
Population: Period 1 mITT population: 54 subjects.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HTD1801 500 mg BID | HTD1801 1000 mg BID | Placebo BID
Number analyzed (Participants) | 15 | 23 | 15
mg/dL | -0.2 (0.52) | 0.0 (0.50) | 0.1 (0.26)

6. Secondary Outcome: Absolute Change in Serum ALP From Week 6 to Week 12 (Period 2)
Time Frame: Week 6 to Week 12
Population: Subjects previously randomized in Period 1 to HTD1801 500 mg BID or HTD1801 1000 mg BID continued for 6 more weeks at that previous dose, while subjects previously randomized to placebo were re-randomized to receive 6 weeks of either HTD1801 500 mg BID or HTD1801 1000 mg BID. 51 subjects in the mITT population started Period 2. 49 subjects in the mITT population completed Period 2.
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- Placebo to HTD1801 500 mg BID: Subjects randomized to receive Placebo BID in Period 1 re-randomized to receive HTD1801 500 mg BID in Period 2
- HTD1801 500 mg BID to HTD1801 500 mg BID: Subjects randomized to receive HTD1801 500 mg BID in Period 1 continuing to receive HTD1801 500 mg BID in Period 2
- Placebo to HTD1801 1000 mg BID: Subjects randomized to receive Placebo BID in Period 1 re-randomized to receive HTD1801 1000 mg BID in Period 2
- HTD1801 1000 mg BID to HTD1801 1000 mg BID: Subjects randomized to receive HTD1801 1000 mg BID in Period 1 continuing to receive HTD1801 1000 mg BID in Period 2
Arm/Group | Placebo to HTD1801 500 mg BID | HTD1801 500 mg BID to HTD1801 500 mg BID | Placebo to HTD1801 1000 mg BID | HTD1801 1000 mg BID to HTD1801 1000 mg BID
Number analyzed (Participants) | 7 | 14 | 7 | 21
U/L | -34 (180.3) | -14 (74.6) | -189 (270.7) | 10 (65.9)

7. Secondary Outcome: Percentage of Subjects Who Achieve ALP of <1.5 x ULN at the End of Week 12 (Period 2)
Time Frame: Week 6 to Week 12
Population: 51 subjects in the mITT population who completed Period 1 and began Period 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo to HTD1801 500 mg BID | HTD1801 500 mg BID to HTD1801 500 mg BID | Placebo to HTD1801 1000 mg BID | HTD1801 1000 mg BID to HTD1801 1000 mg BID
Number analyzed (Participants) | 7 | 15 | 7 | 22
Participants | 0 | 2 | 0 | 6

8. Secondary Outcome: Percentage of Patients Who Achieve a 50% Decrease in ALP at the End of Week 12 (Period 2)
Time Frame: Week 6 to Week 12
Population: 51 subjects in the mITT population who completed Period 1 and began Period 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo to HTD1801 500 mg BID | HTD1801 500 mg BID to HTD1801 500 mg BID | Placebo to HTD1801 1000 mg BID | HTD1801 1000 mg BID to HTD1801 1000 mg BID
Number analyzed (Participants) | 7 | 15 | 7 | 22
Participants | 1 | 0 | 0 | 2

9. Secondary Outcome: Percentage of Patients Who Normalize ALP at the End of Week 12 (Period 2)
Time Frame: Week 6 to Week 12
Population: 51 subjects in the mITT population who completed Period 1 and began Period 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo to HTD1801 500 mg BID | HTD1801 500 mg BID to HTD1801 500 mg BID | Placebo to HTD1801 1000 mg BID | HTD1801 1000 mg BID to HTD1801 1000 mg BID
Number analyzed (Participants) | 7 | 15 | 7 | 22
Participants | 0 | 0 | 0 | 2

10. Secondary Outcome: Absolute Change in Serum Total Bilirubin at the End of Week 12 (Period 2)
Time Frame: Week 6 to Week 12
Population: 49 subjects in the mITT population who completed Period 2.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo to HTD1801 500 mg BID | HTD1801 500 mg BID to HTD1801 500 mg BID | Placebo to HTD1801 1000 mg BID | HTD1801 1000 mg BID to HTD1801 1000 mg BID
Number analyzed (Participants) | 7 | 14 | 7 | 21
mg/dL | -0.1 (0.28) | 0.0 (0.25) | -0.4 (0.16) | 0.0 (0.49)

11. Secondary Outcome: Absolute Change in Serum ALP From Week 12 to Week 18 (Period 3)
Description: Change in serum ALP between a new baseline at Week 12 and the final value at Week 18 for all subjects following the randomized withdrawal
Time Frame: Week 12 to Week 18
Population: All subjects were re-randomized to either continue on the active treatment they received in Period 2 or be assigned to placebo. 50 subjects in the mITT population started Period 3. 49 subjects in the mITT population completed Period 3.
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- HTD1801 500 mg BID to HTD1801 500 mg BID: Subjects who received 500 mg HTD1801 BID in Period 2 re-randomized to continue receiving HTD1801 500 mg BID in Period 3.
- HTD1801 1000 mg BID to HTD1801 1000 mg BID: Subjects who received 1000 mg HTD1801 BID in Period 2 re-randomized to continue receiving HTD1801 1000 mg BID in Period 3.
- HTD1801 500 mg BID to Placebo: Subjects who received 500 mg HTD1801 BID in Period 2 re-randomized to receive Placebo in Period 3.
- HTD1801 1000 mg BID to Placebo: Subjects who received 1000 mg HTD1801 BID in Period 2 re-randomized to receive Placebo in Period 3.
Arm/Group | HTD1801 500 mg BID to HTD1801 500 mg BID | HTD1801 1000 mg BID to HTD1801 1000 mg BID | HTD1801 500 mg BID to Placebo | HTD1801 1000 mg BID to Placebo
Number analyzed (Participants) | 9 | 14 | 12 | 14
U/L | -63 (88.9) | 21 (141.7) | 183 (292.0) | 142 (163.7)

12. Secondary Outcome: Percentage of Patients Who Achieve ALP of <1.5 x ULN at the End of Week 18 (Period 3)
Description: The percentage of patients who achieve ALP of <1.5 x ULN at the end of week 18 (Period 3)
Time Frame: Week 12 to Week 18
Population: 50 subjects in the mITT population who completed Period 2 and began Period 3.
Measure: Count of Participants; unit: Participants
Arm/Group | HTD1801 500 mg BID to HTD1801 500 mg BID | HTD1801 1000 mg BID to HTD1801 1000 mg BID | HTD1801 500 mg BID to Placebo | HTD1801 1000 mg BID to Placebo
Number analyzed (Participants) | 10 | 14 | 12 | 14
Participants | 1 | 4 | 0 | 1

13. Secondary Outcome: Percentage of Patients Who Achieve a 50% Decrease in ALP at the End of Week 18 (Period 3)
Time Frame: Week 12 to Week 18
Population: 50 subjects in the mITT population who completed Period 2 and began Period 3.
Measure: Count of Participants; unit: Participants
Arm/Group | HTD1801 500 mg BID to HTD1801 500 mg BID | HTD1801 1000 mg BID to HTD1801 1000 mg BID | HTD1801 500 mg BID to Placebo | HTD1801 1000 mg BID to Placebo
Number analyzed (Participants) | 10 | 14 | 12 | 14
Participants | 1 | 0 | 0 | 1

14. Secondary Outcome: Percentage of Subjects Who Normalize ALP at the End of Week 18 (Period 3)
Time Frame: Week 12 to Week 18
Population: 50 subjects in the mITT population who completed Period 2 and began Period 3.
Measure: Count of Participants; unit: Participants
Arm/Group | HTD1801 500 mg BID to HTD1801 500 mg BID | HTD1801 1000 mg BID to HTD1801 1000 mg BID | HTD1801 500 mg BID to Placebo | HTD1801 1000 mg BID to Placebo
Number analyzed (Participants) | 10 | 14 | 12 | 14
Participants | 0 | 1 | 0 | 0

15. Secondary Outcome: Absolute Change in Serum Total Bilirubin at the End of Week 18 (Period 3)
Time Frame: Week 12 to Week 18
Population: 49 subjects in the mITT population who completed Period 3.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HTD1801 500 mg BID to HTD1801 500 mg BID | HTD1801 1000 mg BID to HTD1801 1000 mg BID | HTD1801 500 mg BID to Placebo | HTD1801 1000 mg BID to Placebo
Number analyzed (Participants) | 9 | 14 | 12 | 14
mg/dL | -0.2 (0.19) | 0.0 (0.23) | 0.1 (0.36) | 0.1 (0.22)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed the informed consent form at the screening date through Study Visit Week 22.
Groups:
- 500mg HTD1801 bid; 1000mg HTD1801 bid: HTD1801: HTD1801 tablets, 250mg
Arm/Group | 500mg HTD1801 bid | 1000mg HTD1801 bid | placebo bid
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/31 | 0/35
Serious Adverse Events (participants affected / at risk) | 1/22 | 3/31 | 0/35
Other Adverse Events (participants affected / at risk) | 14/22 | 20/31 | 18/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 500mg HTD1801 bid (N=22) | 1000mg HTD1801 bid (N=31) | placebo bid (N=35)
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 500mg HTD1801 bid (N=22) | 1000mg HTD1801 bid (N=31) | placebo bid (N=35)
Diarrhoea (Gastrointestinal disorders) | 0 | 7 | 0
Nausea (Gastrointestinal disorders) | 0 | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0
Inflammatory Bowel Disease (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 3 | 2
Upper Respiratory Tract Infection (Gastrointestinal disorders) | 0 | 2 | 1
Sinusitis (Gastrointestinal disorders) | 1 | 0 | 1
Bronchitis (Gastrointestinal disorders) | 0 | 0 | 1
Clostridium Difficile Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Cystitis (Gastrointestinal disorders) | 0 | 1 | 0
Influenza (Gastrointestinal disorders) | 1 | 0 | 0
Laryngitis (Gastrointestinal disorders) | 0 | 1 | 0
Localised Infection (Gastrointestinal disorders) | 0 | 1 | 0
Oral Herpes (Gastrointestinal disorders) | 0 | 1 | 0
Tonsillitis (Gastrointestinal disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 5 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hair Texture Abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Spider Naevus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 5
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 3
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 3
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 0 | 3
Liver Function Test Increased (Investigations) | 0 | 0 | 3
Blood Bilirubin Increased (Investigations) | 0 | 1 | 1
Blood Potassium Decreased (Investigations) | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 2 | 1
Influenza Like Illness (General disorders) | 2 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 0
Chest Pain (General disorders) | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 1
Cervical Radiculopathy (Nervous system disorders) | 1 | 0 | 0
Lumbar Radiculopathy (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sputum Increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal Column Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Stoma Site Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0
Hot Flush (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT03333928/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/28/NCT03333928/SAP_001.pdf